CLINICAL TRIAL: NCT04131530
Title: Automatic Evaluation of Inflammation Activity in Ulcerative Colitis Using Probe-based Confocal Laser Endomicroscopy With Artificial Intelligence
Brief Title: Automatic Evaluation of Inflammation Activity in Ulcerative Colitis Using pCLE With Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of QiLu Hospital, Shandong University
Other Study IDs: 2019SDU-QILU-10
Record Dates: First submitted 2019-10-17; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Ulcerative Colitis; Artificial Intelligence; Confocal Laser Endomicroscopy
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopist will observe the colon mucosa of UC using pCLE and take biopsy for histology examination.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colon mucosa observed by pCLE: pCLE is used to evaluate the inflammation activity in different parts of the colon mucosa
  Interventions: Diagnostic Test: The diagnosis of Artificial Intelligence and endoscopist

INTERVENTIONS:
Diagnostic Test: The diagnosis of Artificial Intelligence and endoscopist — When the colon mucosa is observed using pCLE, endoscopist and AI will make a diagnosis independently. In addition, the endoscopist can not see the diagnosis of AI.

SUMMARY:
Probe-based confocal laser endomicroscopy (pCLE) is an endoscopic technique that enables to evaluate the inflammation activity of ulcerative colitis with excellent correlation with histopathology. However this requires much experience, which limits the application of pCLE. The investigators designed a computer-aided diagnosis program using deep neural network to make diagnosis automatically in pCLE examination and contrast its performance with endoscopists.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80; diagnosed as UC

Exclusion Criteria:

* Patients under conditions unsuitable for performing CLE including coagulopathy , impaired renal or hepatic function, pregnancy or breastfeeding, and known allergy to fluorescein sodium; Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the endoscopy pCLE examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The diagnosis efficiency of Artificial Intelligence | 3 months
  The primary outcome is to test the diagnostic accuracy, sensitivity, specificity, PPV, NPV of the Artificial Intelligence for evaluation of inflammation activity of UC on pCLE examination.

SECONDARY OUTCOMES:
Contrast the diagnosis efficiency of Artificial Intelligence with endoscopists | 3 months
  The secondary outcome is to compare the diagnosis efficiency (including diagnostic accuracy, sensitivity, specificity, PPV, NPV ) between Artificial Intelligence and endoscopists.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China